CLINICAL TRIAL: NCT06790784
Title: A Randomized Clinical Trial Evaluating Combination Faricimab + PRP vs. Vitrectomy + Endolaser for Treatment of Proliferative Diabetic Retinopathy
Brief Title: Faricimab + PRP vs. Vitrectomy + Endolaser for Treatment of PDR
Acronym: AP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol AP; UG1EY014231 (NIH)
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Proliferative Diabetic Retinopathy (PDR)
Keywords: faricimab; vitrectomy; endolaser; panretinal photocoagulation
MeSH Terms: interventions — Vitrectomy; faricimab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Faricimab + PRP (Experimental): PRP = Panretinal Photocoagulation
  Interventions: Drug: Faricimab; Device: Panretinal Photocoagulation (PRP)
- Vitrectomy + Endolaser (Active Comparator)
  Interventions: Procedure: Vitrectomy; Device: Endolaser

INTERVENTIONS:
Procedure: Vitrectomy — The vitrectomy must occur within 4 weeks of randomization. A single injection of faricimab is allowed at any point before the vitrectomy. It is recommended that this injection is within 1 week of the vitrectomy. Requirement of triamcinolone staining to assist in complete elevation and removal of the posterior hyaloid and in removal of as much peripheral vitreous as is safely possible, 20 gauge not permitted. Allows subconjunctival steroid at investigator discretion; however, sub-tenon's triamcinolone or other long-acting steroid will not be permitted.
  Arms: Vitrectomy + Endolaser
Device: Endolaser — Complete panretinal photocoagulation (PRP) during vitrectomy
  Arms: Vitrectomy + Endolaser
Drug: Faricimab — Treatment must be initiated on the day of randomization with one faricumab injection. The remainder of the randomized treatment includes 2 additional injections every 4-weeks. Injections must be completed within 90 days of randomization.
  Arms: Faricimab + PRP
Device: Panretinal Photocoagulation (PRP) — Complete PRP. PRP may be completed in 1-3 sessions, with the timing at the investigator's discretion. All PRP sessions must be completed within 90 days of randomization.
  Arms: Faricimab + PRP

SUMMARY:
This randomized trial will compare treatment strategies for proliferative diabetic retinopathy (PDR). Participants will receive either combination a of faricimab + PRP or vitrectomy + endolaser. The participants will be followed for 3 years. The study will evaluate long-term visual acuity as well as differences in number of injections, procedures, and complications during follow-up (after completion of randomization treatment), and cost.

DETAILED DESCRIPTION:
Although some combination of anti-VEGF plus PRP is the most common treatment approach for PDR with and without DME, there are currently no long-term data on a standardized approach. Vitrectomy is not currently used as first-line treatment for early PDR but advances in surgical technique have reduced associated complications and the ability to remove the posterior hyaloid during surgery may have advantages over nonsurgical approaches, especially in the reduction of vitreous hemorrhage and/or traction retinal detachment that may occur later when the hyaloid separates naturally. Protocol S demonstrated both PRP and anti-VEGF alone result in good visual acuity results long-term so it is expected that a combination treatment would also result in good visual acuity results.

This study will evaluate the safety and efficacy of two treatment strategies for PDR: faricimab plus PRP and Vitrectomy with endolaser with the goal to determine whether either approach decreases visit and treatment burden along with decreasing complications compared with the other treatment method while maintaining good visual acuity. The primary objectives of this study are to compare visual acuity at 3 years following vitrectomy with endolaser or faricimab+PRP and to compare number of treatments for PDR (i.e., injections, PRP, vitrectomy) following the end of randomized treatment over 3 years.

ELIGIBILITY:
Inclusion Criteria:

Individual:

* ≥ 18 years old
* Diagnosis of diabetes mellitus (type 1 or type 2)

Study Eye:(A participant can have one or two study eyes if both eyes are eligible at screening.)

* Presence of PDR requiring treatment, defined as moderate PDR or worse on global grading of ultrawide field fundus photos or NV meeting criteria for moderate PDR or worse on global grading of ultrawide field FA, confirmed by a central reading center
* Best corrected visual acuity ≥49 letters (20/100 Snellen equivalent or better)

Exclusion Criteria:

* Individual:

  * Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
  * Blood pressure > 160/100 (systolic above 160 or diastolic above 100).

    o If blood pressure is brought below 160/100 by anti-hypertensive treatment, individual can become eligible.
  * For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.

    * Women of childbearing potential will be required to have pregnancy testing or use an acceptable method of pregnancy prevention. Women who are potential study participants should be questioned about the potential for pregnancy at baseline and prior to each injection. Pregnancy test is required for all women of childbearing potential at baseline. Investigator judgment is used to determine when a pregnancy test is needed during follow up.

Study Eye: (A participant can have two study eyes.)

* Traction retinal detachment involving the macula
* Significant vitreous hemorrhage that would preclude completion of a full PRP
* Significant vitreomacular traction
* Any prior vitrectomy
* Any prior PRP (defined as ≥100 burns outside of the posterior pole)
* Treatment for DME within the prior 6 months
* Intravitreal anti-VEGF for any indication, other than DME, within the prior year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2031-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity Change from Baseline | Baseline to 3- years
  Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40.
Number of Post-Randomization Treatments for Proliferative Diabetic Retinopathy | Over 3 Years
  Initial randomized treatment will be excluded.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Retina Associates of Southern California, Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - Florida Retina Consultants, Lakeland, Florida
  - Ophthalmic Partners of Florida, PA dba Central Florida Retina, Orlando, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Illinois Retina Associates SC Oak Park Site, Oak Park, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Wolfe Clinic, P.C.- West Des Moines, West Des Moines, Iowa
  - Mid-America Retina Consultants, P.A., Overland, Kansas
  - University of Kentucky Advanced Eye Care, Lexington, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Boston Medical Center Corporation, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Retina Research Institute, LLC, St Louis, Missouri
  - Retina Associates of Western NY, P.C., Rochester, New York
  - Retina-Vitreous Consultants, Inc., Monroeville, Pennsylvania
  - Retina Consultants of Texas, PA, Bellaire, Texas
  - Texas Retina Associates, Lubbock, Texas